CLINICAL TRIAL: NCT03739931
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study of mRNA-2752, a Lipid Nanoparticle Encapsulating mRNAs Encoding Human OX40L, IL-23, and IL-36γ, for Intratumoral Injection Alone and in Combination With Immune Checkpoint Blockade
Brief Title: Dose Escalation Study of mRNA-2752 for Intratumoral Injection to Participants in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-2752-P101; 2022-001597-55 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dose Escalation: Relapsed/Refractory Solid Tumor Malignancies or Lymphoma; Dose Expansion: Triple Negative Breast Cancer, HNSCC, Non-Hodgkins, Urothelial Cancer, Immune Checkpoint Refractory Melanoma, and NSCLC Lymphoma
Keywords: mRNA-2752; OX40L; IL-23; IL-36γ; Intratumoral injection
MeSH Terms: conditions — Lymphoma; Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: mRNA-2752 (Experimental): Participants will be administered mRNA-2752 at an applicable dose as monotherapy.
  Interventions: Biological: mRNA-2752
- Arm B: mRNA-2752 + Durvalumab (Experimental): Participants will be administered mRNA-2752 at an applicable dose in combination with durvalumab.
  Interventions: Biological: mRNA-2752; Biological: Durvalumab
- Arm C: mRNA-2752 Alone or mRNA-2752 + Durvalumab (Experimental): Participants will be administered mRNA-2752 at an applicable dose as monotherapy or in combination with durvalumab.
  Interventions: Biological: mRNA-2752; Biological: Durvalumab

INTERVENTIONS:
Biological: mRNA-2752 — Solution for intratumoral injection
Biological: Durvalumab — Solution for infusion after dilution
  Arms: Arm B: mRNA-2752 + Durvalumab; Arm C: mRNA-2752 Alone or mRNA-2752 + Durvalumab

SUMMARY:
The clinical study will assess the safety and tolerability of escalating intratumoral doses of mRNA-2752 in participants with relapsed/refractory solid tumor malignancies or lymphoma.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter, dose-escalation study of intratumoral injections of mRNA-2752 alone and in combination with intravenously administered immune checkpoint blockade therapy in participants with histologically confirmed advanced or metastatic solid tumor malignancies or lymphoma. The study consists of Dose Escalation and Dose Confirmation Parts, which will occur in Arm A and Arm B, followed by a Dose Expansion Part, which will occur in Arm B, and a Dose Exploration in Arm C as a neoadjuvant therapy for cutaneous melanoma.

Participants in Arm A and in Arm B will be enrolled into the Dose Escalation Part and the doses of mRNA-2752 will be administered in a dose escalation regimen until a maximum tolerated dose (MTD) or a recommended dose for expansion (RDE) is identified. When the MTD/RDE is identified, participants with solid tumors or lymphoma with visceral lesions may be enrolled into the Dose Confirmation Part to confirm that the dose is also appropriate for this subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to completing any study-specific procedure
* Histologically confirmed advanced or metastatic disease with at least 1 measurable lesion as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Cheson 2016 criteria
* Dose Escalation/Confirmation:

  o Has disease progression after adequate standard of care therapies for metastatic disease that are known to confer clinical benefit, is intolerant to treatment, or refuses standard treatment (no limit to prior lines of therapy)
* Dose Expansion:

  * Group 1 Triple negative breast cancer: Must have objective evidence of disease progression during or following at least one prior line of therapy for metastatic or locally advanced disease. Enrollment to Stage 3 of this cohort will include participants who have previously progressed on prior immune checkpoint blockade or participants with programmed death-ligand 1 (PD-L1) negative tumor based on archival tissue (if available).
  * Group 2 Head and neck squamous cell carcinoma: Must have objective evidence of disease progression during or following platinum-containing chemotherapy as well as a PD-1/L1 therapy
  * Group 3 Non-Hodgkin's lymphoma: Must have objective evidence of disease progression and have received 2 or more prior lines of therapy. Participants with large B-cell lymphoma must have received prior anthracycline containing chemotherapy.
  * Group 4 Urothelial cancer, first line: Must be cisplatin ineligible and PD-L1 negative
  * Group 5 Urothelial cancer: Must have objective evidence of disease progression during or following platinum-containing chemotherapy
  * Group 6 Cutaneous melanoma: Must be refractory to immune checkpoint blockade in the primary or secondary acquired resistance setting.
  * Group 7 Non-small cell lung cancer, primary refractory or secondary acquired resistance to immune checkpoint blockade.
* Dose Exploration:

  o Newly diagnosed resectable, BRAF wild-type, Stage IIIB/C/D and Stage IV cutaneous melanoma with clinically evident lymph node involvement in the neoadjuvant setting.
* Has a tumor lesion amenable to biopsy and must be willing to provide the baseline and on-treatment tumor biopsy samples if medically feasible. For participants with only 1 lesion amenable to injection, biopsy, and RECIST assessment, that lesion must be ≥2 centimeters (cm)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
* Has a body weight of >30 kilograms (kg)
* Adequate hematological and biological function
* Has evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants
* Treatment Arm B and Arm C: Clinical euthyroid status. Participants with clinically stable hypothyroidism, on adequate thyroid supplementation, are permitted on study.

Exclusion Criteria:

* Has received prior systemic anticancer therapy including investigational agents within 5 half-lives or 28 days of the start of study treatment, whichever is shorter. Participants enrolled to Arm C may not have received any previous anti-cancer therapy, immune therapy, radiotherapy, or investigational agents.
* Has received prior radiotherapy within 14 days before the first dose of study treatment. Participants enrolled to Arm C may not have had prior anticancer therapy including radiotherapy.
* Has received a live vaccine within 30 days before the first dose of study treatment
* Has current or prior use of immunosuppressive medication within 14 days before the first dose of study treatment
* Have major surgical procedures within 28 days or non-study-related minor procedures within 7 days before the first dose of study treatment.
* Requires active systemic anticoagulation at the time of intratumoral injection or biopsy
* Active central nervous system tumors or metastases
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and protocol defined laboratory values

  * Participants with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Medical Monitor.
  * Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Medical Monitor.
* Any active or prior documented autoimmune or inflammatory disorders
* History of primary immunodeficiency, allogenic solid organ transplantation, or tuberculosis
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the participant to give written informed consent
* Has active GI bleeding or hemoptysis or history of bleeding disorder
* Is a female participant who is pregnant or breastfeeding or male or female participant of reproductive potential who are not willing to employ effective birth control from screening to 120 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to Day 28
Number of Participants with Adverse Events (AEs) | Up to 27 months
Arm B: Overall Response Rate (ORR): Percentage of Participants with Tumor Response (Partial or Complete) Based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) in Cutaneous Melanoma | Up to 2 years

SECONDARY OUTCOMES:
ORR: Percentage of Participants with Tumor Response (Partial or Complete) Based on RECIST v1.1 and modified RECIST (iRECIST), and Cheson and Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) for Participants With Lymphoma | Up to 2 years
Pharmacokinetics: Maximum Observed Concentration (Cmax) | Predose, immediately after injection, and 15 minutes up to 168 hours postdose

CONTACTS AND LOCATIONS:
Locations (24):
- United States (16):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Providence St. John's Health Center, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Sarasota, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cancer Center at Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Australia (4):
  - One Clinical Research Perth, Nedlands, Western Australia
  - Alfred Health, Melbourne
  - Westmead Hospital, Westmead
  - Melanoma Institute of Australia, Wollstonecraft
- Israel (4):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srikrishna D, Sachsenmeier K. We need to bring R0 < 1 to treat cancer too. Genome Med. 2021 Jul 26;13(1):120. doi: 10.1186/s13073-021-00940-9. PMID 34311780